CLINICAL TRIAL: NCT00359879
Title: Safety and Efficacy of Exenatide Taken Before Lunch and Before Dinner Compared With Before Breakfast and Before Dinner in Patients With Type 2 Diabetes Using Oral Antidiabetic Therapy
Brief Title: Comparison of Exenatide Taken Before Lunch and Dinner With Before Breakfast and Dinner in Patients With Type 2 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H8O-CR-GWBH
Record Dates: First submitted 2006-08-01; First posted 2006-08-03 (Estimated); Last update posted 2015-02-23 (Estimated); Status verified 2015-01

CONDITIONS: Type 2 Diabetes
Keywords: diabetes; exenatide; Lilly; Amylin
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Exenatide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 - exenatide before breakfast and dinner (Experimental)
  Interventions: Drug: exenatide
- 2 - exenatide before lunch and dinner (Active Comparator)
  Interventions: Drug: exenatide

INTERVENTIONS:
Drug: exenatide — subcutaneous injection, 5mcg or 10mcg, twice a day (before lunch and dinner)
  Other Names: Byetta
  Arms: 2 - exenatide before lunch and dinner
Drug: exenatide — subcutaneous injection, 5mcg or 10mcg, twice a day (before breakfast and dinner)
  Other Names: Byetta
  Arms: 1 - exenatide before breakfast and dinner

SUMMARY:
This trial is designed to compare the effects of twice-daily (before lunch and before dinner) exenatide plus oral antidiabetic (OAD) agents and twice-daily (before breakfast and before dinner) exenatide plus OAD with respect to glycemic control (HbA1c) in patients with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with type 2 diabetes.
* Have been treated with one of the following treatment regimens for at least three months prior to screening: *metformin alone; *sulfonylurea (SU) alone; *thiazolidinedione (TZD) alone; *a combination of metformin and SU; *a combination of metformin and TZD.
* HbA1c between 7.1% and 10.0%, inclusive.
* Body Mass Index (BMI) > 25 kg/m^2 and < 45 kg/m^2

Exclusion Criteria:

* Have participated in an interventional, medical, surgical, or pharmaceutical study (a study in which an experimental drug, medical, or surgical treatment was given) within 30 days prior to screening.
* Have characteristics contraindicating metformin, SU, or TZD use.
* Are receiving chronic (lasting longer than 2 weeks) systemic glucocorticoid therapy (excluding topical and inhaled preparations) or have received such therapy within 2 weeks immediately prior to screening.
* Have used any prescription drug to promote weight loss within 3 months prior to screening.
* Are currently treated (for greater than 2 consecutive weeks) with any of the following excluded medications: *insulin within 3 months prior to screening; *alpha-glucosidase inhibitors within 3 months prior to screening; *meglitinides within 3 months prior to screening; *drugs that directly affect gastrointestinal motility

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 377 (Actual)
Dates: Start 2006-09; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Change in HbA1c (glycosylated hemoglobin) from Baseline to Week 12 | Baseline, Week 12
  Evaluate the change in glycemic control as measured by HbA1c from Baseline to Week 12

SECONDARY OUTCOMES:
Change in body weight from Baseline to Week 12, and if measured, at each visit | Baseline, Weeks 4, 8, 12
  Change in body weight (kg) from Baseline to Week 12, and if measured, at each visit in between (Weeks 4 and 8)
Change in fasting serum glucose (FGS) from Baseline to Week 12, and if measured, at each visit | Baseline, Weeks 4, 8, 12
  Change in FGS from Baseline to Week 12, and if measured, at each visit in between (Weeks 4 and 8)
Changes in self-monitored blood glucose (SMBG) profile from Baseline through Week 12 | Baseline, Weeks 4, 8, 12
  Changes in glucose measured at different times throughout the day derived from 7-point SMBG profile (glucose measurements before and 2 hours after the start of the morning, midday, and evening meals, and at bedtime)

CONTACTS AND LOCATIONS:
Overall Officials: James Malone, MD, Study Director — Eli Lilly and Company
Locations (15):
- Brazil (9):
  - Research Site, Campinas
  - Research Site, Curitiba
  - Research Site, Fortaleza
  - Research Site, Goiânia
  - Research Site, Porto Alegre
  - Research Site, Rio de Janeiro
  - Research Site, Salvador
  - Research Site, São José do Rio Preto
  - Research Site, São Paulo
- Mexico (6):
  - Research Site, Aguascalientes, Aguascalientes
  - Research Site, Guadalajara, Jalisco
  - Research Site, Monterrey, Nuevo León
  - Research Site, San Luis Potosí City, San Luis Potosí
  - Research Site, Mérida, Yucatán
  - Research Site, Mexico City

REFERENCES:
- [Derived] Forti A, Garcia EG, Yu MB, Jimenez MC, Brodows RG, Oliveira JH. Efficacy and safety of exenatide administered before the two largest daily meals of Latin American patients with type 2 diabetes. Curr Med Res Opin. 2008 Sep;24(9):2437-47. doi: 10.1185/03007990802282398. Epub 2008 Jul 24. PMID 18662495